CLINICAL TRIAL: NCT06172894
Title: An Open-label, Multi-center, Dose-escalation Phase Ib Study to Determine the Recommended Phase 2 Dose of APN401 in Patients with Advanced Solid Tumors
Brief Title: PBMC-based Leukocyte Immunotherapy
Acronym: PALINDROM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: invIOs GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APN401-104
Record Dates: First submitted 2023-11-24; First posted 2023-12-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
Keywords: ATMP (Advanced Therapy Medicinal Product); PBMCs (Peripheral Blood Mononuclear Cells); Cbl-b (Casitas B Lineage Lymphoma B); advanced solid tumor; siRNA (small interfering ribonucleic acid); cell therapy; immune checkpoint

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APN401 (Experimental): Intravenous infusion of APN401 in 3-weekly (i.e. 21 days) intervals for a maximum of 4 doses at either 1.5x10^7 PBMCs/kg (i.e., Dose Level 1) or 4.5x10^7 PBMCs/kg (i.e., Dose Level 2), depending on assigned cohort
  Interventions: Drug: APN401

INTERVENTIONS:
Drug: APN401 — APN401 is a suspension of viable peripheral blood mononuclear cells (PBMCs) from an individual patient that have been transfected with a small interfering ribonucleic acid (siRNA) to reduce Cbl-b expression. It is administered intravenously in 3-weekly intervals (i.e. every 21 days) for a maximum of 4 treatment cycles.

SUMMARY:
This is an open-label, multicenter, dose-escalation Phase Ib trial of APN401, a suspension of viable Peripheral Blood Mononuclear Cells (PBMCs) from an individual patient that have been transfected with a small interfering ribonucleic acid (siRNA) to reduce Cbl-b expression. Twelve evaluable participants with advanced solid tumors will be assessed. The primary objective is to evaluate the safety and tolerability of APN401 and to determine the Recommended Phase 2 Dose (RP2D) of APN401. The secondary objective is to collect preliminary data on the clinical efficacy of APN401.

Participants will receive up to four APN401 treatments via intravenous infusion at 3-weekly intervals. Participants, who have completed four treatment cycles and a safety follow-up, will be contacted by telephone to evaluate survival status at 6 and 12 months after start of treatment.

DETAILED DESCRIPTION:
APN401 is a suspension of autologous Peripheral Blood Mononuclear Cells (PBMCs), transiently transfected with an siRNA to reduce Cbl-b protein levels. The administration of autologous Cbl-b silenced PBMCs to the patient will promote activation of both adaptive and innate immune mechanisms targeting tumor cells; along these lines APN401 is assumed to demonstrate significant improvement in cancer immune therapy. In addition, silencing of Cbl-b in the context of cellular therapeutics has potential to reduce mortality rates for patients with advanced cancers.

This is an open-label, single-arm trial to be conducted with up to twelve patients at four hospitals in Austria, Europe. Two dose levels of APN401 are evaluated using a Bayesian Optimal Interval (BOIN) study design with accelerated titration:

* Dose Level/Cohort 1: 1.5x10^7 PBMCs/kg
* Dose Level/Cohort 2: 4.5x10^7 PBMCs/kg

Dose escalation requires at least one patient to be treated and observed for at least three weeks after the first dose. The BOIN method will be used to guide the dose level assignment and estimate the MTD/RP2D based on cumulative information on DLTs in Cycle 1 of treatment (i.e. 3 weeks after first dose).

Patients with advanced solid tumors first undergo screening procedures during a 28-day time window between giving consent and starting APN401 treatment. Eligible patients are treated with up to four APN401 infusions. During each treatment cycle, patients undergo leukapheresis on the first day and APN401 infusion on the second day (i.e., D0/D1; D21/D22; D42/D43; D63/D64). During the subsequent follow-up phase, patients participate a safety-follow up 3 weeks post last APN401 dose and are contacted by telephone to evaluate survival status at 6 and 12 months after start of treatment. Tumor imagings to evaluate the efficacy of APN401 treatment are scheduled during the screening phase (baseline imaging), and prior to treatment Cycle 3 and the last Safety Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 18 years or older (all genders)
2. Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors and who have failed standard treatment, have no standard treatment, or are not suitable for standard treatment at this stage as determined by the investigator
3. Progressed on or refractory to at least two prior lines of systemic therapy
4. At least one measurable lesion according to RECIST 1.1
5. An Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
6. Life expectancy of at least 3 months
7. Adequate organ and bone marrow function, in the absence of growth factors, defined by specific laboratory parameters.
8. Negative serology for human immunodeficiency virus, syphilis, hepatitis B and hepatitis C
9. No prior chemotherapy, radiation therapy (except for palliative purpose), endocrine therapy, immunotherapy or investigational agent within 3 weeks (or five half-lives) prior to Day 0 (6 weeks for nitrosoureas and mitomycin C) before treatment
10. Toxicities from previous anti-cancer therapies or surgical procedures to grade ≤1 that have not resolved (except alopecia)
11. Previous exposure to a checkpoint inhibitor is allowed (except exposure of Cbl-b inhibition)
12. Women of childbearing potential must have a negative pregnancy test, should not be breastfeeding, and must be willing to use highly effective methods of contraception for at least 1 month before, while participating in this study and until 1 month after the end of the treatment
13. Patient voluntarily agrees to participate in this study and signs an Ethics Committee approved informed consent prior to performing any of the screening visit procedures, indicating that the patient understands the purpose and procedures required for the study
14. Patient is not participating in any other interventional clinical study within the past 30 days

Exclusion Criteria:

1. Active untreated brain metastases
2. Use of systemic corticosteroids (> 10 mg prednisone or equivalent) within 15 days (except for prophylaxis for radiodiagnostic contrast reactions), or other immunosuppressive drugs within 30 days, prior to the first dose of APN401. Replacement therapy (e.g., physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
3. Active, known, or suspected autoimmune disease except type I diabetes, vitiligo and thyroid disorders (thyroxine or insulin replacement therapy is allowed)
4. Patients at high medical risk because of non-malignant systemic disease, active or unstable cardiac or cerebro-vascular disease, or active uncontrolled infection
5. Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or APN401 administration, or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the patient unsuitable for the study
6. Any vaccination prior and/or after 7 days while on APN401 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) and/or Serious Adverse Events (SAEs) | Up to 30 days post last dose
  The safety and tolerability of APN401 will be assessed by recording the TEAEs and SAEs using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0)
Occurence of Dose Limiting Toxicities (DLTs) | Observed from Day 1 of APN401 infusion until the end of Cycle 1 (Day 21)
  The safety and tolerability of APN401 will be assessed by recording DLTs
Determination of Recommended Phase 2 Dose (RP2D) of APN401 | Through completion of DLT period of last evaluable patient, an average of 8 months
  RP2D will be determined on the BOIN recommendations (based on DLT and MTD) and the overall safety information

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 months
  Preliminary data on clinical efficacy of APN401 will be assessed according to RECIST 1.1
Disease Control Rate (DCR) | Up to 12 months
  Preliminary data on clinical efficacy of APN401 will be assessed according to RECIST 1.1
Overall Survival (OS) | Time from enrollment to death
  Preliminary data on clinical efficacy of APN401 will be assessed
Overall Survival (OS) at 3, 6 and 12 months | At 3, 6 and 12 months post start of treatment phase
  Preliminary data on clinical efficacy of APN401 will be assessed
Progression Free Survival (PFS) | From date of enrollment until the date of first evidence of disease progression or date of death from any cause, whichever came first, assessed up to 12 months
  Preliminary data on clinical efficacy of APN401 will be assessed according to RECIST 1.1
Progression Free Survival (PFS) Rate at 3 months | At 3 months post start of treatment phase
  Preliminary data on clinical efficacy of APN401 will be assessed according to RECIST 1.1
Immune responses in circulation to monitor APN401 immune activation | Prior to treatment cycles C1, C2, C3, C4 (each cycle is 21 +/- 3 days) and 21 days (+/-10 days) post last APN401 dose
  Preliminary data on clinical efficacy of APN401 will be assessed using ELISA-based techniques

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (4):
  - Salzburg Cancer Research Institute (SCRI), Center for Clinical Cancer and Immunology Trials (CCCIT), Salzburg, Salzburg
  - Medizinische Universität Innsbruck, Universitätsklinik für Innere Medizin V, Hämatologie und internistische Onkologie, Innsbruck, Tyrol
  - Ordensklinikum Linz, Barmherzige Schwestern, Abteilung für Hals-, Nasen-, Ohrenheilkunde, Linz, Upper Austria
  - Medizinische Universität Wien, Universitätsklinik für Transfusionsmedizin und Zelltherapie, Vienna, Vienna